CLINICAL TRIAL: NCT04284995
Title: A Phase 2 Open Label Study to Assess the PK and PD Properties of a Single Subcutaneous Injection of RUC-4 in Patients With a ST-elevation Myocardial Infarction Presenting to the Cardiac Catheterization Lab With Planned Primary Coronary Angioplasty
Brief Title: A Phase 2 Open Label Study to Assess the PK/PD Properties of RUC-4 in Patients With a ST-elevation Myocardial Infarction
Acronym: CEL-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CeleCor Therapeutics (Industry)
Collaborators: St. Antonius Hospital (Other); Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CEL-02
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Coronary Disease; Myocardial Infarction; Heart Diseases; Vascular Diseases; STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; Myocardial Infarction; Heart Diseases; Vascular Diseases; ST Elevation Myocardial Infarction | interventions — RUC-4 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): Cohort 1: 0.075 mg/kg RUC-4. 8 STEMI Patients will be enrolled.
  Interventions: Drug: RUC-4 Compound
- Cohort 2 (Experimental): Cohort 2: Dose of RUC-4 selected by Safety Review Committee (SRC) after completion of Cohort 2 and review of data. 8 STEMI Patients will be enrolled.
  Interventions: Drug: RUC-4 Compound
- Cohort 3 (Experimental): Cohort 3: Dose of RUC-4 selected by Safety Review Committee (SRC) after completion of Cohort 2 and review of data. 8 STEMI Patients will be enrolled.
  Interventions: Drug: RUC-4 Compound

INTERVENTIONS:
Drug: RUC-4 Compound — All patients will receive a single subcutaneous dose of RUC-4 in the Cardiac Catheterization Lab (CCL) before coronary angiography/percutaneous coronary intervention.

SUMMARY:
RUC-4 is a novel, promising and fast acting (5-15 minutes) αIIbβ3 receptor antagonist with a high-grade inhibition of platelet aggregation (≥80%) shortly after subcutaneous administration. This study is designed to extend the findings in CEL-01 to patients with ST-elevation myocardial Infarction (STEMI) presenting to the cardiac catheterization laboratory with planned coronary angioplasty.

DETAILED DESCRIPTION:
RUC-4 is a novel, promising and fast acting (5-15 minutes) αIIbβ3 receptor antagonist with a high-grade inhibition of platelet aggregation (≥80%) shortly after subcutaneous administration. For patients with ST-elevation myocardial infarction (STEMI) early treatment with RUC-4 could be beneficial by improving initial patency of the infarct related vessel and by minimizing thrombotic occlusions, thus improving both coronary artery and myocardial microvascular blood flow, possibly resulting in a decrease in infarct size and a reduction in complications of STEMI.

The purpose of this study is to assess the PD and PK properties of a single subcutaneous injection of RUC-4 in STEMI patients presenting to the cardiac catheterization laboratory with planned coronary angioplasty. In addition the safety and tolerability will be assessed at baseline and hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI, presenting with persistent chest pain (>30 min) and ≥1 mm ST-segment elevation in two adjacent electrocardiograph leads, with >6 mm cumulative ST-segment deviation, in whom the total duration of symptoms to first intracoronary device deployment (excluding a wire) is anticipated to be within 6 hours
2. Adult males and females 18 years of age or older
3. Females must be non-pregnant, non-lactating, and of non-childbearing potential (postmenopausal or surgically sterilized) by history and review of medical record
4. Weight (by history) of between 52 and 120 kg
5. Written informed consent (following short-form of the informed consent form at Cardiac Catheterization Lab)

Exclusion Criteria:

1. High probability in the opinion of the cardiologist that current STEMI is caused by stent thrombosis and the previous PCI related to this stent thrombosis is <1 month
2. High suspicion of type II MI
3. Out of hospital cardiac arrest (OHCA)
4. Therapy resistant cardiogenic shock (systolic blood pressure ≤80 mm Hg for >30 minutes)
5. Persistent severe hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg)
6. Current active coronavirus disease 2019 (COVID-19) infection (criteria according to local guidelines)
7. Known severe liver disease
8. Known history of severe renal dysfunction (glomerular filtration rate <30 mL/min or serum creatinine >200 mmol/L [>2.5 mg/dL])
9. Known left bundle branch block
10. Requirement of oral anticoagulation (Vitamin K antagonists {VKA} or direct oral antagonists {DOACs})
11. Current treatment with αIIbβ3 receptor antagonist (other than RUC-4)
12. Coagulation abnormality, known bleeding disorder, or history of documented prior hemorrhagic or thrombotic stroke within the past 6 months
13. History of upper or lower GI bleeding within the past 6 months
14. Known clinically important anemia
15. Known clinically important thrombocytopenia (platelet count of less than 150,000/μL)
16. Known history of allergy to any of the ingredients in the RUC-4 formulation (i.e., acetate buffer, sucrose)
17. Major surgery within the past 6 months
18. Life expectancy of less than 6 months
19. Any clinically significant abnormality identified prior to enrollment that in the judgment of the Investigator would preclude safe completion of the study
20. Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the patient's ability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Platelet Inhibition | Baseline
  Inhibition of Platelet Aggregation
Platelet Inhibition | 15 minutes
  Inhibition of Platelet aggregation
Platelet inhibition | 45 minutes
  Inhibition of Platelet aggregation
Platelet inhibition | 60 minutes
  Inhibition of Platelet aggregation
Platelet inhibition | 90 minutes
  Inhibition of Platelet aggregation
Platelet inhibition | 120 minutes
  Inhibition of Platelet aggregation
Platelet inhibition | 180 minutes
  Inhibition of Platelet aggregation
RUC-4 Concentration | Baseline
  concentration in blood (ng/mL)
RUC-4 Concentration | 15 minutes
  concentration in blood (ng/mL)
RUC-4 Concentration | 45 minutes
  concentration in blood (ng/mL)
RUC-4 Concentration | 90 minutes
  concentration in blood (ng/mL)
RUC-4 Concentration | 120 minutes
  concentration in blood (ng/mL)
RUC-4 Concentration | 180 minutes
  concentration in blood (ng/mL)
Safety and Tolerability | Baseline
  Bleeding events, Injection site reactions,vital signs, ECG, laboratory results
Safety and Tolerability | Hospital discharge
  Bleeding events, Injection site reactions,vital signs, ECG, laboratory results
RUC-4 Concentration | 240 minutes
  concentration in blood (ng/mL)
Platelet aggregation | 240 minutes
  Inhibition of platelet aggregation

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius hospital, Nieuwegein, CM, Netherlands

IPD SHARING:
Plan to Share IPD: No